CLINICAL TRIAL: NCT06022796
Title: Weight Loss Interventions for Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202300165
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Overweight; Weight Loss; Ketogenic Dieting; Obesity
MeSH Terms: conditions — Overweight; Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial, participants in the HK-RTE group will be advised to follow a healthy ketogenic diet with RTE meals provided (n=25), with a maximum of 50g net carbohydrate intake daily. Those in the control group will be instructed to follow a healthy ketogenic diet (HKD) (n=25).
Masking Description: It is not feasible to apply blinding to the study design due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Ketogenic Ready-To-Eat (HK-RTE) Meals (Experimental): Participants in the HK-RTE group (n=25) will be provided with the Healthfull meals for lunch and dinner in the first month. They will be advised to take these meals as part of a healthy ketogenic diet, with a maximum of 50g total net carbohydrates daily.
  Participants will receive nutrition education conducted by dietitians over the course of 6 months (total of 5 dietary workshops covering topics such as ketogenic dietary advice and self-monitoring habits). Participants will also receive health coaching via the Nutritionist Buddy (nBuddy) mobile application to facilitate monitoring of diet intake, physical activity and weight throughout the 6 months study period.
  Interventions: Other: Healthy Ketogenic Ready-to-Eat Meals
- Healthy Ketogenic Diet (HKD) (Active Comparator): Participants in the reference group will be instructed to follow a Healthy Ketogenic Diet (n = 25), with a maximum of 50g total net carbohydrates daily.
  Similar to the experimental group, participants will receive nutrition education conducted by dietitians over the course of 6 months (total of 5 dietary workshops such as ketogenic dietary advice and self-monitoring habit). Participants will also receive health coaching via the Nutritionist Buddy (nBuddy) mobile application to facilitate monitoring of diet intake, physical activity and weight throughout the 6 months study period.
  Interventions: Other: Healthy Ketogenic Diet

INTERVENTIONS:
Other: Healthy Ketogenic Ready-to-Eat Meals — Participants will be provided nutrition education via 5 dietary workshops focusing on a healthy ketogenic diet. In addition, HK-RTE meals will be provided to participants as a form of meal replacement for lunch and dinner over 1 month. Participants will be expected to follow a healthy ketogenic diet thereafter.
  Other Names: Very low carbohydrate diet
  Arms: Healthy Ketogenic Ready-To-Eat (HK-RTE) Meals
Other: Healthy Ketogenic Diet — Participants will receive nutrition education via 5 dietary workshops focusing on a healthy ketogenic diet, without the provision of HK-RTE meals.
  Arms: Healthy Ketogenic Diet (HKD)

SUMMARY:
Numerous barriers towards weight management among Singaporeans with obesity exists, which involves environmental and self-regulation factors (i.e. motivation and hunger). Hence, the provision of healthy ketogenic ready-to-eat meals may be a potential solution to facilitate initial weight loss through increasing motivation while reducing appetite and hunger levels among these individuals. Therefore, this study will investigate the effect of healthy ketogenic ready-to-eat meals with mHealth nutrition application versus healthy ketogenic diet (without meal provision) with the mHealth nutrition app to facilitate weight loss and improve metabolic outcomes among individuals with obesity.

DETAILED DESCRIPTION:
In Singapore, the widespread availability of local meals and concerns of overconsumption due to a lack of internal self-regulation skills for hunger predisposes an increased energy intake. Furthermore, a lack of time, motivation, and self-efficacy in preparing healthy meals may potentially limit the extent of weight and dietary management among local individuals with obesity.

The ketogenic diet has consistently demonstrated beneficial effects on facilitating weight management. This weight loss mechanism involves achieving a calorie deficit, induced state of nutritional ketosis, and the reduction in appetite and hunger. Importantly, the weight loss achieved from the early phase of the intervention serves as one of the key enablers in the weight loss process. Despite these benefits, there is paucity in the literature examining the provision of healthy ketogenic ready-to-eat (HK-RTE) meals on weight loss. Furthermore, none of these studies explored the extent of motivation derived from the benefits of these meals, nor included the use of mHealth self-monitoring strategies to encourage weight loss.

To address the research gap, our study aims to evaluate the effectiveness of HK-RTE meals with mHealth app, as compared to healthy ketogenic diet (HKD) (without meal provision) using the mHealth app on weight loss and metabolic outcomes among Asian individuals with obesity.

In this randomized controlled trial, participants will be randomized to either HK-RTE group or the HKD group using computer-generated random sequencing. Both groups will receive nutrition education conducted by dietitians throughout the 6-month study period (total of 5 dietary workshops covering topics such as ketogenic dietary advice and self-monitoring habits).

The HK-RTE group will be provided with HK-RTE meals for lunch and dinner in the first month (n = 25). They are to take these meals as part of a healthy ketogenic diet, with a maximum of 50g net total carbohydrates daily. Those in the control group will be advised to follow a healthy ketogenic diet (HKD) without the RTE meals (n = 25) and similarly to keep to a maximum of 50g net carbohydrates daily. Participants will also be encouraged to use the Nutritionist Buddy (nBuddy) mobile application to facilitate monitoring of diet intake, physical activity and weight throughout the 6-month study period. The impact of the HK-RTE meals on motivation and appetite regulation in influencing weight loss will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 75 years old
* Body Mass Index >= 27.5kg/m2
* Own a smartphone
* Literacy in English
* NUH staff

Exclusion Criteria:

* Intention of pregnancy; Pregnancy; Lactating individuals
* Type 1 Diabetes Mellitus or Type 2 Diabetes Mellitus on insulin treatment
* Untreated Endocrinopathy (e.g., hyper/hypothyroidism)
* Advanced kidney disease
* Abnormal liver function test assessed at screening
* Heart diseases
* Severe cognitive or psychiatric disabilities/disorders (e.g., eating disorders, depression)
* Active malignancies
* Taking medications that affect appetite or induce weight loss; previous or plans for bariatric surgery.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | 1 month, 3 months, 6 months
  Weight changes post-intervention

SECONDARY OUTCOMES:
Blood pressure | 3 months, 6 months
  Systolic and diastolic changes at follow up appointments
Hemoglobin A1c | 3 months, 6 months
  HbA1c changes at follow up appointments
Fasting blood glucose | 3 months, 6 months
  Fasting blood glucose changes at follow up appointments
Total cholesterol | 3 months, 6 months
  Cholesterol changes at follow up appointments
Low-density lipoprotein cholesterol | 3 months, 6 months
  Cholesterol changes at follow up appointments
High-density lipoprotein cholesterol | 3 months, 6 months
  Cholesterol changes at follow-up appointments
Triglycerides | 3 months, 6 months
  Triglycerides changes at follow up appointments
Motivation to initiate and maintain dietary behaviours | 3 months, 6 months
  Motivation via self-reported questionnaire
Perceived competence to maintain dietary behaviour | 3 months, 6 months
  Perceived competence via self-reported questionnaire
Hunger | 3 months, 6 months
  Subjective ratings of hunger feelings via self-reported questionnaire
Dietary intake | 6 months
  Nutrients intake by assessing food logs in nBuddy application

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore